CLINICAL TRIAL: NCT03839108
Title: Which is More Effective: Prolotherapy or Paraffin Waxes for Hand Ostearthritis
Brief Title: Comparison of Effect of Prolotherapy and Paraffin Waxes for Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Işıl Üstün, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/419
Record Dates: First submitted 2019-02-05; First posted 2019-02-15 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hand Osteoarthritis
Keywords: paraffin; prolotherapy; hand osteoarthritis
MeSH Terms: interventions — Paraffin; Prolotherapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: randomised single blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin wax group (Active Comparator): Paraffin group patients will be told to take of jewellery and dip their hands into the bath of melted wax (52 ºC) with hands open and hand wrist in neutral position for 10 times .In paraffin wax group, patients will be treated 5 days a week for 2 weeks period. Paraffin wax bath will be applied for 20 minutes in every physical therapy session.
  Interventions: Other: Paraffin wax
- Prolotherapy group (Experimental): Drug = prolotherapy (%15 dextrose solution) into hand joints
  %15 dextrose solution will be injected into medial and lateral aspect of proximal interphalangeal joints (PIJ), distal interphalangeal joints and carpometacarpal joint of thumb for 3 sessions once a week period.
  Interventions: Drug: Prolotherapy

INTERVENTIONS:
Other: Paraffin wax — Paraffin group patients will be told to take of jewellery and dip their hands into the bath of melted wax (52 ºC) with hands open and hand wrist in neutral position for 10 times .In paraffin wax group, patients will be treated 5 days a week for 2 weeks period. Paraffin wax bath will be applied for 20 minutes in every physical therapy session.
  Other Names: paraffin
  Arms: Paraffin wax group
Drug: Prolotherapy — . Prolotherapy is a nonsurgical regenerative injection technique that introduces small amounts of an irritant solution to the site of painful and degenerated tendon insertions (entheses), joints, ligaments, and in adjacent joint spaces during several treatment sessions to promote growth of normal cells and tissues.Hypertonic dextrose solution is most common used agent. In prolotheraphy group, %15 dextrose solution will be applied to medial and lateral aspect of proximal interphalangeal joints (PIJ), distal interphalangeal joints and carpometacarpal joint of thumb for 3 sessions once a week period
  Arms: Prolotherapy group

SUMMARY:
Patients with hand osteoarthritis will be randomized into two groups, paraffin wax and prolotherapy group. Patients will be evaluated before and after treatment , after 2 weeks 4 weeks and 3 months after treatment. Evaluation parameters are visual analog scale, Duruoz hand index scales, grip strength, lateral pinch, two point pinch and three point pinch strengths.

DETAILED DESCRIPTION:
This study is a randomized clinical trial. 40 Patients with hand osteoarthritis will be randomized into 2 groups, paraffin wax and prolotherapy group.Paraffin group patients will be told to take of jewellery and dip their hands into the bath of melted wax (52 ºC) with hands open and hand wrist in neutral position for 10 times .In paraffin wax group, patients will be treated 5 days a week for 2 weeks period. Paraffin wax bath will be applied for 20 minutes in every physical therapy session. Prolotherapy is a nonsurgical regenerative injection technique that introduces small amounts of an irritant solution to the site of painful and degenerated tendon insertions (entheses), joints, ligaments, and in adjacent joint spaces during several treatment sessions to promote growth of normal cells and tissues.Hypertonic dextrose solution is most common used agent. In prolotherapy group, %15 dextrose solution will be applied to medial and lateral aspect of proximal interphalangeal joints (PIJ), distal interphalangeal joints and carpometacarpal joint of thumb for 3 sessions once a week period. Grip strength, lateral pinch, two point pinch, three point pinch strengths, Visual analog scale (VAS), Duruoz Hand Index scales will be assessed before the intervention and after two weeks, 4 weeks and 3 months after intervention .

ELIGIBILITY:
Inclusion Criteria:

* Hand osteoarthritis defined according to American College of Rheumatology criteria
* Older than 40 years

Exclusion Criteria:

* Carpal tunnel syndrome
* De quervain tenosynovitis
* Dupuytren's contracture
* Secondary osteoarthritis due to Rheumatoid arthritis, chondrocalcinosis, Psoriatic arthritis, hemachromatosis
* Trigger finger

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Changed pain score >%20 in hand osteoarthritis in paraffin wax group measured by Visual Analog Scale at 3 months | 3 months
  Pain is measured by visual analog scale (VAS). The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm). The patients' pain in paraffin wax group are assessed by VAS in 3 months. Changed pain score >%20 VAS is one of the primary outcomes
Changed pain score >%20 in hand osteoarthritis in prolotherapy group measured by Visual Analogue Scale | 3 months
  pain change is measured by Visual analogue scales (VAS). The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm). Changed pain score >%20 VAS in prolotherapy group are assessed in 3 months.
Comparison of effect of prolotherapy and paraffin wax on pain score change | 3 months
  VAS score changes of two groups will be compared

SECONDARY OUTCOMES:
Duruoz Hand Index Scale | 3 months
  The DHI is a self-report questionnaire which was developed about 15 years ago to evaluate the capacity to carry out manual functional activities with no assistance or aids in patients with rheumatoid arthritis .
  It consists of 18 questions regarding manual tasks which are frequently carried out while cooking, washing, dressing, etc. The patient is asked to evaluate the difficulty which he/she has in carrying out these tasks (from 0: no difficulty, to 4: nearly impossible)
  The psychometric properties of this scale have been evaluated in patients with rheumatoid arthritis, scleroderma, hand osteoarthritis, stroke, trauma , diabetes and patients on haemodialysis. Duruoz Hand Index Scales of both groups before the treatment, 3 months after treatment will be compared
Grip strength, lateral pinch strength, three point strength, two point pinch strength | 3 months
  Grip strength, lateral pinch strength, three point strength, two point pinch strength is measured by dynamometer in both groups before and after treatment. Effect of therapy on strength of hands will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Işıl Üstün, Principal Investigator — Bakırköy Dr. Sadi Konuk Training and Research Hospital; Sibel Çağlar Okur, Study Director — Dr Sadi Konuk Training and Research Hospital
Locations (1):
- University of Health Sciences Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results of the study will be written as a manuscript. In Turkey, we do not have a system sharing data to other researchers

REFERENCES:
- [Background] Dilek B, Gozum M, Sahin E, Baydar M, Ergor G, El O, Bircan C, Gulbahar S. Efficacy of paraffin bath therapy in hand osteoarthritis: a single-blinded randomized controlled trial. Arch Phys Med Rehabil. 2013 Apr;94(4):642-9. doi: 10.1016/j.apmr.2012.11.024. Epub 2012 Nov 24. PMID 23187044
- [Background] Jahangiri A, Moghaddam FR, Najafi S. Hypertonic dextrose versus corticosteroid local injection for the treatment of osteoarthritis in the first carpometacarpal joint: a double-blind randomized clinical trial. J Orthop Sci. 2014 Sep;19(5):737-43. doi: 10.1007/s00776-014-0587-2. Epub 2014 Aug 27. PMID 25158896